CLINICAL TRIAL: NCT01095367
Title: Seprafilm™ for the Prevention of Intraperitoneal Adhesions and Improved Delivery of Therapy in Women Undergoing Staging and Intraperitoneal Chemotherapy for Advanced Ovarian Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to company changes and lack of funding-unlikely to have sufficient numbers to analyze meaningfully
Sponsor: University of British Columbia (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H09-03436
Record Dates: First submitted 2010-03-22; First posted 2010-03-30 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Adhesion barrier sheets; ovarian cancer; Advanced stage epithelial ovarian cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms | interventions — Seprafilm

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Seprafilm™ (Active Comparator): Subject will have 3 sheets of Seprafilm™ placed in her abdominal cavity (in the pelvis, upper abdomen and below the incision) at the end of debulking surgery. At 7-21 days after surgery the subject will receive a contrast dye, Iohexol (Omnipaque™), into her intraperitoneal port. The subject will then undergo 3 abdominal X-rays, to assess the extent of abdominal adhesions.
  Interventions: Procedure: Seprafilm™
- No Seprafilm™ (No Intervention): Subject will undergo debulking surgery without Seprafilm™ placement (standard care). At 7-21 days after surgery the subject will receive a contrast dye, Iohexol (Omnipaque™), into her intraperitoneal port. The subject will then undergo 3 abdominal X-rays, to assess the extent of abdominal adhesions.

INTERVENTIONS:
Procedure: Seprafilm™ — Seprafilm™ Adhesion Barrier is an approved temporary, bioresorbable adhesion barrier to reduce the incidence, extent, and severity of adhesions in patients undergoing abdominal or pelvic laparotomy.
  Seprafilm sheets are size 5" x 6" individually-wrapped, sterile membranes. Three or more Seprafilm™ sheets will be placed in the randomized cohort.
  Other Names: Adhesion Barrier sheets
  Arms: Seprafilm™

SUMMARY:
The purpose of this research is to determine if a film to prevent adhesions will improve the area of distribution of a contrast dye (representative of chemotherapy) in the abdominal cavity (belly) of women who have undergone surgery for ovarian cancer as compared with patients who have not had adhesion barrier sheets placed in the belly. It is believed that this film, Seprafilm™, reduces adhesions (scar tissue between tissues and organs) in the abdominal cavity following surgery. Adhesions can limit the distribution of the chemotherapy agent placed in the abdomen to treat the ovarian cancer. Thirty subjects will receive adhesion barrier sheets and thirty will not. To determine if the sheets prevent adhesions, all subjects will have a dye inserted into the abdomen and then have X-rays of the abdomen to look at the distribution of the dye between the two groups.

Hypothesis:

Null hypothesis: There is no difference in area of distribution of the intraperitoneal dye in the Seprafilm ™ vs. no Seprafilm™ groups.

Alternative hypothesis: Seprafilm™ reduces adhesion formation and there is a larger area of distribution of intraperitoneal dye in the Seprafilm™ group.

DETAILED DESCRIPTION:
The recommended treatment of epithelial ovarian cancer (EOC) includes optimal surgical debulking to < 1 cm residual disease, followed by a combination of intraperitoneal (IP) and intravenous (IV) chemotherapy for at least 6 cycles. Serous EOC is known to spread transperitoneally and is often diffusely disseminated within the peritoneal cavity. It is believed that IP therapy via direct contact is effective in treating such small intraperitoneal implants. What is not known is whether IP therapy is evenly distributed in individuals and to what degree adhesions and formation of scar tissue prevents the even distribution of chemotherapy within the belly, potentially impacting efficacy. Few studies have addressed the question of adhesions and intraperitoneal therapy in general, and there have been no studies specifically in ovarian cancer utilizing current guidelines. Efficacy has been proven for IP/IV therapy over IV alone but the range of survival within the IP group may be secondary to "tumor biology," patient selection (i.e., disease truly > 1 cm) or lack of/poor distribution of IP drug secondary to adhesions. Any product that could be shown to decrease those adhesions and increase the area of distribution of IP therapy would prove a major advantage.

The majority of scarring and adhesions take place in the first 7 days after a surgical procedure. And the first IP and IV chemotherapy usually commences between 7-21 days after surgery. Therefore, the first treatment provides an opportunity to assess intraperitoneal adhesions. To assess adhesions, we will inject radiopaque dye (iohexol) via the IP port, rotate the patient per the standard practice during IP therapy to distribute the injected liquid, and then take 3 views (simple X-rays) of the abdomen. The area of distribution of the dye (representing distribution of IP chemotherapy) will be compared in two groups of subjects (Seprafilm™ vs. no Seprafilm™).

ELIGIBILITY:
Inclusion Criteria:

* Epithelial ovarian cancer
* Stage III or IV (advanced)
* Planned intraperitoneal chemotherapy
* Optimally debulked to less than 1 cm residual tumor in any area within the peritoneal cavity (after consent prior to randomization)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-04; Primary Completion 2012-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The area of distribution of contrast dye in the intraperitoneal cavity as measured on three abdominal films taken 7-10 days following debulking surgery for epithelial ovarian cancer. | 7-10 days

SECONDARY OUTCOMES:
The safety and side effects of placement of Seprafilm, including fever, elevated WBC count, nausea, blocked port, port infection, small bowel obstruction
The safety and side effects of IP omnipaque dye injection, including fever, elevated WBC count, nausea, blocked port, port infection, small bowel obstruction
The additional time taken for 1) placement of Seprafilm, 2) injection of IP contrast dye, 3) obtaining 3-way abdominal X-rays, and 4) interpretation of films

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Dianne Miller, Study Director — British Columbia Cancer Agency; Mark S Carey, MD, Study Director — University of British Columbia; Thomas G Ehlen, MD, Study Director — University of British Columbia; Sarah Finlayson, MD, Principal Investigator — University of British Columbia; Janice Kwon, MD, Study Director — University of British Columbia; Gavin CE Stuart, MD, Study Director — University of British Columbia; Anna Tinker, MD, Study Director — British Columbia Cancer Agency; Mark Heywood, MD, Study Director — University of British Columbia
Locations (2):
- University of Nevada School of Medicine, Las Vegas, Nevada, United States
- Vancouver General Hospital, Vancouver, British Columbia, Canada